CLINICAL TRIAL: NCT02871466
Title: Intra Cardiac Autologous Stem Cells Infusion May Improve Clinical Outcomes in Failing Heart Subjects Refractory to Maximal Drug Therapy and Internal Cardioverter With a Defibrillator (ICD) Recipients
Brief Title: Stem Cells Therapy in Advanced Heart Failure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, principal investigator, University of Campania Luigi Vanvitelli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8.2016
Record Dates: First submitted 2016-08-10; First posted 2016-08-18 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stem cells infusion (Experimental)
  Interventions: Drug: stem cells infusion

INTERVENTIONS:
Drug: stem cells infusion

SUMMARY:
stem cells therapy may be a choice therapy for advanced heart failure patients refractory to medical therapy, internal cardiovertor with a defibrillator (ICD) recipients, and a previous history of myocardial infarction and coronary artery revascularization. These patients, without indication to receive a cardiac resynchronization therapy (CRT), may have a worsening of heart failure, and symptoms of coronary artery disease. In this study we have evaluated in consecutive 30 selected patients the amelioration in failing heart NYHA class, hospitalization rate, echocardiographic left ventricle functionality, and associated to reduction of angina after a treatment with stem cells intra thoracic infusion.

ELIGIBILITY:
Inclusion Criteria:

* heart failure post coronary artery disease, refractory to maximal medical therapy, previous coronary artery surgical revascularization.

Exclusion Criteria:

* inflammatory chronic diseases, neoplastic diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-01; Primary Completion 2022-01 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
NYHA class improvement | 12 months
reduction in hospitalization rate | 12 months
reduction in angor symptoms | 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Celestino Sardu, Naples
  - Raffaele Marfella, Naples
  - Celestino Sardu, Napoli

IPD SHARING:
Plan to Share IPD: No